CLINICAL TRIAL: NCT04787003
Title: A Single-arm, Open-label Clinical Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of Oncolytic Virus (OVV-01) Injection Combined With or Without Immune Checkpoint Inhibitors in the Treatment of Patients With Advanced Solid Tumors
Brief Title: Oncolytic Virus (OVV-01) Injection in the Treatment of Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: North China Petroleum Bureau General Hospital (Other)
Collaborators: Joint Biosciences Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RR-001
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Neoplasms
Keywords: Oncolytic Virus Injection; Intratumoral Injection; Immune Checkpoint Inhibitors
MeSH Terms: conditions — Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncolytic virus (OVV-01) injection for patients with advanced solid tumors (Experimental): Oncolytic virus (OVV-01) injection combined with or without immune checkpoint inhibitors in the treatment of patients with advanced solid tumors.
  Interventions: Drug: oncolytic virus (OVV-01) injection

INTERVENTIONS:
Drug: oncolytic virus (OVV-01) injection — intratumoral injection of OVV-01 with or without immune checkpoint inhibitors
  Other Names: C045

SUMMARY:
Phase Ia: To investigate the safety, tolerability and efficacy of OVV-01 injection in the treatment of patients with advanced solid tumors (OVV-01 single dose gradient exploration).

Phase Ib: To evaluate the safety, tolerability and efficacy of OVV-01 injection combined with immune checkpoint inhibitors pembrolizumab (anti-PD-1 monoclonal antibody) or atezolizumab (anti-PD-L1 monoclonal antibody) in the treatment of patients with advanced solid tumors (OVV-01 combined with PD-1/PD-L1 monoclonal antibody dose gradient exploration);

Phase Ic: A cohort expansion of Phase Ib to further analyze the efficacy and safety of OVV-01 injection combined with immune checkpoint inhibitor injection in the treatment of advanced solid tumors.

DETAILED DESCRIPTION:
Phase Ia:

This is a prospective, multicenter, open-label, single-arm investigator-initiated clinical study to evaluate the safety and efficacy of intratumoral injection of OVV-01 injection in patients with advanced solid tumors.

This study plans to enroll in 1 ~ 3 study sites nationwide about 9 ~ 18 patients with advanced solid tumors for whom the standard treatment failed and currently no standard treatment is available or standard treatment is not suitable due to medical reasons, to conduct a phase Ia study, i.e., the First in Human (FIH) trial of OVV-01 injection, using the traditional "3 + 3" approach for dose gradient exploration.

Phase Ib:

This is a prospective, multi-center, open-label, single-arm investigator-initiated clinical study to evaluate the safety and efficacy of intratumoral injection of OVV-01 injection combined with immune checkpoint inhibitors in patients with advanced solid tumors.

This study plans to enroll in 1 ~ 3 study sites nationwide about 12 ~ 24 patients with advanced solid tumors for whom the standard treatment failed and currently no standard treatment is available or standard treatment is not suitable due to medical reasons, to conduct a phase Ib study, using the traditional "3 + 3" approach and based on the phase Ia results, 2 dose gradients of OVV-01 are used in combination with pembrolizumab and atezolizumab, respectively, to explore the efficacy and safety.

Phase Ic:

This is a prospective, multi-center, open-label, single-arm investigator-initiated clinical study to evaluate the safety and efficacy of intratumoral injection of OVV-01 injection combined with immune checkpoint inhibitors in patients with advanced solid tumors.

This study plans to enroll in 1 ~ 3 study sites nationwide about 15 ~ 20 patients with advanced solid tumors for whom the standard treatment failed and currently no standard treatment is available or standard treatment is not suitable due to medical reasons, to conduct a phase Ic study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 and ≤ 70 years;
2. Patients with advanced solid tumors confirmed by histopathological/cytological examination of the primary tumor and/or metastases, including but not limited to: melanoma, head and neck squamous cell carcinoma, cervical cancer, osteosarcoma, nasopharyngeal carcinoma, breast cancer, lung cancer, colorectal cancer, liver cancer, gastric cancer;
3. Patients for the third-line or higher standard therapy failed;
4. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (non-nodal lesions with longest diameter ≥ 10 mm, or nodal lesions with short diameter ≥ 15 mm);
5. ECOG score of 0 ~ 2;
6. Expected survival ≥ 3 months;
7. Adequate bone marrow function;

   * WBC ≥ 3.0 × 109/L;
   * Neutrophils (ANC) ≥ 1.5 × 109/L;

     Lymphocyte count ≥ 6.0 × 108/L
   * Platelets ≥ 90 × 109/L without transfusion within 14 days prior to starting the first cell therapy;
   * Hemoglobin ≥ 10.0 g/dL
8. Adequate hepatic and renal function:

   Total bilirubin ≤ 1.5 × ULN.
   * AST and ALT < 2.5 × ULN; < 5 × ULN AST for patients with liver metastases;
   * Blood creatinine ≤ 1.5 × ULN, or creatinine clearance rate ≥ 50 ml/min (calculation with Cockcroft/Gault formula)
9. Coagulation function:

   * INR ≤ 1.5 × ULN
   * PTT ≤ 1.5 × ULN
10. Adequate cardiovascular function:

    * Epilepsy score (EF) ≥ 50%
    * QTcF interval ≤ 450 ms
11. Women of childbearing age who have a negative pregnancy test within 14 days before treatment. Female patients of childbearing age, and male patients with partners of childbearing age must agree to use at least one medically recognized contraceptive method (such as surgical sterilization, oral contraceptives, intrauterine device, sexual abstinence or barrier contraception combined with spermicide, etc.) during study treatment and within at least 6 months after the last dose of investigational drug;
12. The patients voluntarily participated in this study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. Subjects without measurable lesions;
2. Subjects with known brain metastasis and/or clinically suspected tumor brain metastasis (patients with asymptomatic brain metastasis or clinically stable for more than 3 months after local treatment can be excluded);
3. Subjects who have received radiotherapy for target lesion within 2 months;
4. Subjects with other active malignancies requiring concurrent treatment;
5. Subjects with known hypersensitivity to the investigational drug or its active ingredients and excipients;
6. Subjects who have received or are still receiving treatment with other investigational drugs or antiviral therapy 4 weeks before randomization;
7. Subjects preparing for or having received tissue/organ transplantation preciously;
8. Subjects having any active infection or unexplained fever > 38.5℃ during the screening period, prior to the first dose;
9. Subjects with active pulmonary tuberculosis (TB) who are receiving anti-TB treatment or who have received anti-TB treatment within 1 year before screening;
10. Subjects with positive result of serological test for Treponema pallidum;
11. Subjects with known positive history of human immunodeficiency virus (HIV) test or known acquired immunodeficiency syndrome (AIDS);
12. Subjects with active hepatitis. Hepatitis B: hepatitis B virus surface antigen (HBVs Ag) positive or HBVsAg negative, but anti-HBVc positive and HBV DNA test value higher than the upper limit of normal; hepatitis C: hepatitis C virus antibody (HCV Ab) positive and HCV RNA positive; with hepatitis B and C co-infection;
13. Cardiovascular system disorders meeting any of the following:

    * Congestive heart failure with cardiac function ≥ NYHA III;
    * Serious arrhythmia requiring medication;
    * Acute myocardial infarction, severe or unstable angina pectoris, coronary artery or peripheral artery bypass grafting or stenting within 6 months prior to the first dose;
    * Left ventricular ejection fraction (LVEF) < 50%;
    * Corrected QTc interval > 450 ms for males and > 470 ms for females, or presence of risk factors for torsades de pointes such as clinically significant hypokalemia, family history of long QT syndrome or family history of arrhythmia (e.g., Wolff-Parkinson-White syndrome) as judged by the investigator;
    * Hypertension not effectively controlled (defined as systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg after standardized antihypertensive drug therapy)
14. Patients with active autoimmune diseases or history of autoimmune diseases that may relapse, but patients with the following diseases are not excluded, may be further screened:

    * Type 1 diabetes;
    * Hypothyroidism (if controlled with hormone replacement therapy alone);
    * Controlled celiac disease;
    * Skin diseases not requiring systemic treatment (e.g., vitiligo, psoriasis, alopecia);
    * Any other disease that will not recur in the absence of external triggers;
15. Patients in any condition requiring systemic treatment with corticosteroids (prednisone > 10 mg/day or equivalent of the similar drug) or other immunosuppressive agents within 14 days prior to investigational drug administration, but currently or previously treated with any of the following steroid regimens, were included:

    * Adrenaline replacement steroid (prednisone ≤ 10 mg/day or equivalent of the similar drug);
    * Topical, ophthalmic, intra-articular, intranasal, or inhaled corticosteroids with minimal systemic absorption;
    * Prophylactic short-term (≤ 7 days) use of corticosteroids (e.g., allergy to contrast media) or for the treatment of non-autoimmune diseases (e.g., delayed hypersensitivity caused by contact allergens);
16. Subjects having mental illness, alcoholism, inability to quit smoking or drug abuse;
17. Female subjects who are pregnant or lactating, or expecting to become pregnant during the trial (from the screening visit until 180 days after dosing) and male subjects who are expecting to father children;
18. Subjects with adverse reactions caused by previous anti-tumor treatment not recovered to (CTCAE 5.0) grade 1 (except alopecia);
19. Subjects having any serious uncontrolled disease or in other conditions that would preclude them from receiving study treatment and are considered unsuitable for this study in the opinion of the investigator.
20. Subjects in other conditions that are considered unsuitable for this study by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
to define the MTD of OVV-01 | 6 months
  to define the maximum tolerated dose (MTD) of intratumoral administration of OVV-01 injection in humans with malignant tumors.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 8 months
  to evaluate the number of Grade III and above side effects assessed by CTCAE v5.0 for patients who received intratumoral administration of OVV-01 injection combined with immune checkpoint inhibitors pembrolizumab (anti-PD-1 monoclonal antibody) or atezolizumab (anti-PD-L1 monoclonal antibody) in patients with advanced solid tumors.

SECONDARY OUTCOMES:
To evaluate the efficacy assessed by the RECISTv1.1 of OVV-01 | 6 months
  to evaluate preliminary efficacy assessed by the RECISTv1.1 of intratumoral administration of OVV-01 injection in the treatment of patients with advanced solid tumors
To evaluate the efficacy assessed by the RECISTv1.1 of OVV-01 with ICIs | 8 months
  to evaluate the preliminary efficacy assessed by the RECISTv1.1 of intratumoral administration of OVV-01 injection combined with immune checkpoint inhibitors pembrolizumab (anti-PD-1 monoclonal antibody) or atezolizumab (anti-PD-L1 monoclonal antibody) in patients with advanced solid tumors

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Lin, Ph.D, Principal Investigator — North China Petroleum Bureau General Hospital
Locations (1):
- North China Petroleum Bureau General Hospital, Cangzhou, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes
After the publication of this study, we could share the IPD. However, this sharing is limited to academic research.
  Person to be contacted: Study Chair-Professor Qiang Lin; Contact information:billhappy001@163.com
Time Frame: After the publication of this study IPD could be shared.The sharing time is set for 5 years
Access Criteria: For the purpose of academic research only

REFERENCES:
- [Derived] Hua Y, Wang C, Li F, Han Y, Zuo D, Lv Y, Sun M, Yuan P, Yuan R, Zhang F, Ma L, Wang Y, Wu H, Zhou G, Lin Q, Wang S, Li N, Lu Y; North China Petroleum Bureau General Hospital. Phase 1, open-label, multicenter, dose escalation safety and tolerability study of oncolytic virus OVV-01 in advanced solid tumors. J Immunother Cancer. 2025 Jun 5;13(6):e011517. doi: 10.1136/jitc-2025-011517. PMID 40480657